CLINICAL TRIAL: NCT05966311
Title: A Multi-center, Feasibility Study to Evaluate the Use and Safety and of the Pediatric PUMA-G System for Percutaneous Ultrasound Gastrostomy
Brief Title: Pediatric Percutaneous Ultrasound Gastrostomy Technique
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: CoapTech (Industry)
Collaborators: Children's Hospital of Philadelphia (Other); Columbia University (Other); Children's National Research Institute (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 220001
Record Dates: First submitted 2023-07-13; First posted 2023-07-28 (Actual); Last update posted 2024-03-29 (Actual); Status verified 2024-03

CONDITIONS: Gastrostomy; Gastrostomy Complications; Pediatric Disorder; Ultrasound
Keywords: Gastrostomy; Pediatric Gastrostomy; Device Feasibility; Device Safety; Ultrasound; POCUS

STUDY DESIGN:
Intervention Model Description: Participants prospectively enrolled are assigned to the interventional treatment procedure using the PUMA-G Peds System. A retrospective comparator is used as a means of comparing outcomes with a similar, historical cohort of patients who received the standard of care treatment procedure.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Percutaneous Ultrasound Gastrostomy (PUG) (Experimental): Enrolled subjects will receive the PUG procedure using the PUMA-G Pediatric System performed by an Interventional Radiologist
  Interventions: Device: Percutaneous Ultrasound Gastrostomy
- Percutaneous Radiologic Gastrostomy (No Intervention): A matched, retrospective control cohort of patients previously admitted to hospital for the placement of gastrostomy tubes by Interventional Radiology will be used to compare performance of the PUMA-G Pediatric System to standard of care.

INTERVENTIONS:
Device: Percutaneous Ultrasound Gastrostomy — Ultrasound guided placement of gastrostomy tube using the PUMA-G Pediatric System
  Other Names: Ultrasound Gastrostomy; PUG; PUMA-G Pediatric Procedure
  Arms: Percutaneous Ultrasound Gastrostomy (PUG)

SUMMARY:
The purpose of this research study is to test a new device called the PUMA-G Pediatric System. The research will measure if the device works well to safely aid doctors placing gastrostomy feeding tubes in children. The PUMA-G Pediatric System is an investigational device that uses ultrasound and magnets to guide insertion of a feeding tube.

DETAILED DESCRIPTION:
This is a multi-center, non-randomized, non-blinded feasibility study to evaluate the performance and safety of the Percutaneous Ultrasound Gastrostomy (PUG) technique in the pediatric population.

A common method for placing gastrostomy tubes currently uses ionizing radiation to aid doctors in procedural steps. Excess radiation usage may present long-term risks to pediatric patients. The PUG procedure, using the PUMA-G Pediatric System, primarily uses ultrasound to guide gastrostomy feeding tube placement.

Up to 40 patients will be enrolled in the study and receive the PUG procedure using the PUMA-G Pediatric System. Following the procedure, patients will be followed during their hospital admission until discharge or up to 30 days. Data will be collected to assess how safe the procedure was and if the procedure used less radiation. Study subjects will be compared to a matched, retrospective cohort of patients who received standard of care gastrostomy tube placement by Interventional Radiology.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent must be obtained from the patient or a Legally Authorized Representative (ex. parent/guardian) before any study-specific assessment is performed
* Weight ≥5 (Phase 0, Phase 1, Phase 2)
* Weight ≥3kg and <10kg (Phase 3)
* Estimated abdominal wall thickness ≤3cm
* Indication for gastrostomy tube placement, with or without jejunal access tubing via gastrostomy tract, determined to be present for any of the following reasons:
* Anatomic: Ear, nose, or throat abnormalities (Pierre-Robin sequence cleft lip palate)
* Neurologic: Head trauma, Cerebral palsy
* Bowel Disease: Short Bowel syndrome, intestinal dysmotility, inflammatory bowel disease, malabsorption
* Failure to Thrive: Cystic Fibrosis, Cholestasis, AID, Chronic renal failure, and food refusal
* Patient determined to be an appropriate candidate for PUG, PEG, or PRG by the clinical care team
* Anticipated discharge > 24 hrs following gastrostomy

Exclusion Criteria:

* Temperature ≥ 38 C
* Systolic BP < 80 or > 180 mmHg
* Heart Rate < 50 or > 160
* Estimated abdominal wall thickness >3cm
* Coagulopathy defined by INR > 1.7 or Platelets <50,000
* Presence of a contraindication to being in proximity to a magnet (e.g. implantable metallic device).
* History of prior gastrostomy, gastrectomy (partial or complete), or abdominal trauma or upper-abdominal surgery.
* Scoliosis
* Atypical organ placement including microgastria
* Involvement in other investigational trials within 30 days prior to screening,
* Pregnant or nursing (lactating) women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive hCG laboratory test
* Patients with HgB < 7g/dL, or fluid resuscitated within 48hrs prior, or received blood transfusion within 48hrs prior, or active life threatening GI bleeding
* Esophageal Diseases: Atresia, stricture, caustic ingestion
* Spinal anomalies or atypical organ placement
* Any other medical condition(s) that may put the patient at risk or influence study results in the investigator's opinion, based on the performance of a pre-procedural assessment.

Ages: 0 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-07-07 (Actual); Primary Completion 2024-08-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
PUMA-G Pediatric System Device-Related Complication Rate | up to 30 days
  A composite rate of the quantity and severity of device related adverse events will be quantified (i.e. linking complications to what are caused by the device) in the post-procedural period including any additional medical/surgical interventions to resolve

SECONDARY OUTCOMES:
Gastrostomy Procedure Complication Rate | up to 30 days
  The rate of other complications during the immediate procedural period between the PUG placement and a historical cohort of matched controls who underwent gastrostomy placement using standard of care Interventional Radiologic gastrostomy tube placement method
Exposure to treatment conditions that pose long term risk to patient health: Ionizing Radiation (Fluoroscopic Time) | up to 30 days
  The quantity of ionizing radiation used during the PUG procedure will be compared to a historical cohort of matched controls who underwent gastrostomy placement using the standard of care Interventional Radiologic gastrostomy tube placement method. Quantities of procedural ionizing radiation will be measured by total fluoroscopic time (min).
Exposure to treatment conditions that pose long term risk to patient health: Ionizing Radiation (Dose Area Product) | up to 30 days
  The quantity of ionizing radiation used during the PUG procedure will be compared to a historical cohort of matched controls who underwent gastrostomy placement using the standard of care Interventional Radiologic gastrostomy tube placement method. Quantities of procedural ionizing radiation will be measured by dose area product (microGy-m2).
Exposure to treatment conditions that pose long term risk to patient health: Ionizing Radiation (Skin Dose) | up to 30 days
  The quantity of ionizing radiation used during the PUG procedure will be compared to a historical cohort of matched controls who underwent gastrostomy placement using the standard of care Interventional Radiologic gastrostomy tube placement method. Quantities of procedural ionizing radiation will be measured by skin dose (mGy).
Exposure to treatment conditions that pose long term risk to patient health: Anesthesia/Sedative Medications | up to 30 days
  The quantity of anesthesia/sedative medications used during the PUG procedure will be compared to a historical cohort of matched controls who underwent gastrostomy placement using the standard of care Interventional Radiologic gastrostomy tube placement method. Medications and total procedural dosages will be quantified.
Exposure to treatment conditions that pose long term risk to patient health: Antibiotic Medications | up to 30 days
  The quantity of antibiotic medications used during the PUG procedure and in the post-procedural timeframe will be compared to a historical cohort of matched controls who underwent gastrostomy placement using the standard of care Interventional Radiologic gastrostomy tube placement method. Medication and dosage will be measured.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Children's National Hospital, Washington D.C., District of Columbia
  - Nyph/Cumc, New York, New York
  - Children's Hospital Of Phildelphia, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No